CLINICAL TRIAL: NCT07397039
Title: The Comparative Efficacy of Focused Extracorporeal Shockwave Therapy and Dry Needling Among Patients With Myofascial Pain Syndrome of the Upper Trapezius Muscle, a Randomized Controlled Trial.
Brief Title: Efficacy of Focused ESWT and Dry Needling Among Patients With Myofascial Pain Syndrome of the Upper Trapezius Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MURA2022/525
Record Dates: First submitted 2022-11-07; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myofascial Pain Syndrome
Keywords: Extracorporeal shockwave therapy, Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focused Extracorporeal Shockwave Therapy (fESWT) (Experimental): The participant will be treated by fESWT plus conservative treatment. fESWT will be applied once a week, for a total of 3 sessions.
  Interventions: Device: Focused Extracorporeal Shockwave Therapy (fESWT)
- Dry needling (DN) (Active Comparator): The participant will be treated by DN plus conservative treatment. DN will be done as a single session.
  Interventions: Other: Dry needling (DN)

INTERVENTIONS:
Device: Focused Extracorporeal Shockwave Therapy (fESWT) — fESWT will be done using an energy flux density of 0.20 - 0.25 millijoule (mJ)/mm2, a frequency of 4 Hz, and 1000 shocks per session which will be done one session per week, for a total of 3 sessions, consecutively.
  Arms: Focused Extracorporeal Shockwave Therapy (fESWT)
Other: Dry needling (DN) — DN will be done by using a sterile technique with a sterile acupuncture needle, a diameter of 0.25 mm, and a length of 30-40 mm.
  The needle will be applied to the painful active trigger point using fan-shaped movements and the fast-in and fast-out technique until the twitching response disappears.
  Arms: Dry needling (DN)

SUMMARY:
Myofascial pain syndrome (MPS) is one of the most common causes of musculoskeletal pain. Among patients with MPS, the upper trapezius muscle appears to be the common muscle that generates pain in the area of upper extremity. The main target treatment for MPS is to eradicate the painful trigger points by using treatment options, such as ultrasound, laser, and dry needling (DN). In the past decade, focused extracorporeal shockwave therapy (fESWT) has become the well-known treatment for pain relief in various musculoskeletal pain conditions. The main advantages of this non-invasive treatment modality are reducing pain, inflammation and promoting tissue healing. However, there were no previous studies compared effects of fESWT to dry needling. Therefore, the present study aims to compare the efficacy of the two treatments in terms of pain reduction and functional improvement.

DETAILED DESCRIPTION:
* This study is a single-blinded non-inferiority randomized controlled trial that will compare the efficacy of fESWT to DN in terms of pain reduction and functional improvement in patients with MPS of the upper trapezius.
* 58 patients will be recruited for the study and randomly allocated to 2 groups, mainly fESWT and DN.
* For the fESWT group, the participants will receive fESWT once a week, for a total of 3 sessions, consecutively. While the participants in the DN group will receive DN at the painful trigger point for 1 session. Moreover, both groups will receive the same conservative treatment, for example, education, exercise, and behavioral modification advice.
* The primary outcome is Visual Analogue Scale (VAS) and the secondary outcomes are Pain Pressure Threshold (PPT) and Neck Disability Index (NDI) which will be recorded at baseline, 1 week, 3 week, and 6 week from baseline.
* Statistical analysis will be performed using Stata to detect statistically significant changes in the same group and differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* The participant who is diagnosed with myofascial pain syndrome based on the criteria listed below:

The trigger point must be in a taut band of the upper trapezius muscle. The trigger point in the muscle is hypersensitivity to pain. Pain radiates to the specific pattern of the upper trapezius muscle. When pressure is applied to the trigger point, the participant perceives the same pain sensation as their pain complaint.

* The participant who has a VAS score of > or = 5 points
* The participant who has had myofascial pain for > or = 3 months

Exclusion Criteria: The participant who has

* Unresolved neurological or musculoskeletal problems, such as fibromyalgia, cervical radiculopathy, and cervical spine fracture.
* History of cervical spine or shoulder surgery
* Uncontrolled underlying diseases, such as psychological problems, cancer, or acute renal or hepatic failure
* Received treatment by other physical modalities or steroid injection into the trigger point within 3 months, or was treated by analgesic drugs within 2 weeks.
* Contraindicated to ESWT or DN
* Refuse to attend the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Changes in VAS were assessed at baseline, and at 4 and 6 weeks following baseline.
  VAS is a subjective tool that is used to measure pain scores. In this study, the 100-numerical scale will be used, in which 0 means "no pain," whereas 100 means "the worst pain." Patients mark the scale to rate the pain score based on their pain perception.

SECONDARY OUTCOMES:
Pain pressure threshold (PPT) | Changes in PPT were assessed at baseline, and at 4 and 6 weeks following baseline.
  PPT is used to assess the strength of a physical stimulus that causes pain. A mechanical pressure is applied over the measured area, such as a muscle. The minimum force that provokes pain is determined as the pain threshold.
The Neck Disability Index (NDI) | Changes in NDI were assessed at baseline and 6 weeks following baseline.
  The Neck Disability Index (NDI) is a self-report questionnaire intended to evaluate patients' disabilities and how much their neck pain impacts their lives. This questionnaire consists of 10 items; 5 points for each item (pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation).

CONTACTS AND LOCATIONS:
Overall Officials: Thitiporn Phakdepiboon, MD, Principal Investigator — Ramathibodi Hospital
Locations (1):
- Ramathibodi Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Desai MJ, Saini V, Saini S. Myofascial pain syndrome: a treatment review. Pain Ther. 2013 Jun;2(1):21-36. doi: 10.1007/s40122-013-0006-y. Epub 2013 Feb 12. PMID 25135034
- [Background] Simplicio CL, Purita J, Murrell W, Santos GS, Dos Santos RG, Lana JFSD. Extracorporeal shock wave therapy mechanisms in musculoskeletal regenerative medicine. J Clin Orthop Trauma. 2020 May;11(Suppl 3):S309-S318. doi: 10.1016/j.jcot.2020.02.004. Epub 2020 Feb 12. PMID 32523286
- [Background] Jun JH, Park GY, Chae CS, Suh DC. The Effect of Extracorporeal Shock Wave Therapy on Pain Intensity and Neck Disability for Patients With Myofascial Pain Syndrome in the Neck and Shoulder: A Meta-Analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2021 Feb 1;100(2):120-129. doi: 10.1097/PHM.0000000000001493. PMID 32520797
- [Background] Park KD, Lee WY, Park MH, Ahn JK, Park Y. High- versus low-energy extracorporeal shock-wave therapy for myofascial pain syndrome of upper trapezius: A prospective randomized single blinded pilot study. Medicine (Baltimore). 2018 Jul;97(28):e11432. doi: 10.1097/MD.0000000000011432. PMID 29995794
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Kinser AM, Sands WA, Stone MH. Reliability and validity of a pressure algometer. J Strength Cond Res. 2009 Jan;23(1):312-4. doi: 10.1519/jsc.0b013e31818f051c. PMID 19130648